CLINICAL TRIAL: NCT03426631
Title: Effect of DAW1033B2 on Obstructive Sleep Apnea
Brief Title: DAW1033B2 in Obstructive Sleep Apnea
Acronym: OsaStimB2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate professor HMS, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014p001033B2
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo before sleep
  Interventions: Drug: Placebo oral capsule
- DAW1033B2 oral capsule (Experimental): DAW1033B2 before sleep
  Interventions: Drug: DAW1033B2 oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo capsule 30 minutes before sleep
  Arms: Placebo
Drug: DAW1033B2 oral capsule — DAW1033B2 capsule 30 minutes before sleep
  Arms: DAW1033B2 oral capsule

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal subjects. In this protocol the investigators will test the effect of DAW1033B2 administered before sleep on OSA phenotype traits and OSA severity during sleep.

ELIGIBILITY:
Inclusion Criterion:

* OSA: AHI > 15

Exclusion Criteria:

* Any medical condition other than well controlled hypertension, diabetes, hyperlipidemia
* Any medication known to influence breathing, sleep/arousal or muscle physiology.
* Claustrophobia.
* Inability to sleep supine.
* Allergy to lidocaine, Oxymetazoline HCl, DAW1033D.
* Individuals with underlying cardiac disease, such as arrhythmias.
* Individuals taking psychiatric medications, or any of the studied medications for medical care.
* History of seizures
* For women: Pregnancy.
* History of panic disorder / hyperventilation syndrome / Attention deficit-hyperactivity disorder (ADHD) / autism

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, DAW1033B2 Second: Placebo-matching DAW1033B2 administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then DAW1033B2 administered 30 mins before normal sleep time on second study night.
- DAW1033B2 First, Placebo Second: DAW1033B2 administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then placebo administered 30 mins before normal sleep time on second study night.
Period: Overall Study
Arm/Group | Placebo First, DAW1033B2 Second | DAW1033B2 First, Placebo Second
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [46.3 to 58.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI, Events/Hour of Sleep)
Description: Based on previous studies the investigators anticipate that DAW1032B2 will reduce AHI more effectively in subjects with moderate sleep apnea, mildly obese (BMI<32), Vpassive > 50% of Veupnea (ventilation during eupneic ventilatory drive)
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: events/hour of sleep
Arm/Group | Placebo | DAW1033B2 Oral Capsule
Number analyzed (Participants) | 12 | 12
events/hour of sleep | 33 [24.1 to 41.9] | 20.4 [6.4 to 47.9]
Statistical Analysis 1: Comparison: Placebo vs DAW1033B2 Oral Capsule; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -11.7

ADVERSE EVENTS:
Time Frame: 1 night
Arm/Group | Placebo | DAW1033B2 Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | DAW1033B2 Oral Capsule (N=12)
Heartburn (gastroesophageal reflux) (Gastrointestinal disorders) | 0 (0) | 1 (1) — The subject referred severe heartburn that resolved after administration of 2 antacid tablets (Calcium 400mg + Sodium 2 mg)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT03426631/Prot_SAP_000.pdf